CLINICAL TRIAL: NCT00465855
Title: Randomized Trial of One Versus Three Hyperbaric Oxygen Treatments for Acute CO Poisoning
Brief Title: One vs. Three Hyperbaric Oxygen Treatments for Acute Carbon Monoxide Poisoning
Acronym: 1V3CORCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Deseret Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1002700
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Carbon Monoxide Poisoning
Keywords: Carbon monoxide poisoning; Hyperbaric oxygen therapy; Randomized controlled trial; Clinical investigation
MeSH Terms: conditions — Carbon Monoxide Poisoning | interventions — Oxyhemoglobins; Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hyperbaric Oxygen (HBO2) - 3 sessions (Active Comparator): Subjects undergo 3 hyperbaric oxygen sessions within 24 hours following carbon monoxide poisoning.
  Interventions: Combination Product: Hyperbaric Oxygen (HBO2) - 3 sessions
- Hyperbaric Oxygen (HBO2) - 1 session (Sham Comparator): Subjects undergo 1 hyperbaric oxygen session and then 2 sham chamber sessions within 24 hours of carbon monoxide poisoning.
  Interventions: Combination Product: Hyperbaric Oxygen (HBO2) - 1 session

INTERVENTIONS:
Combination Product: Hyperbaric Oxygen (HBO2) - 3 sessions — Before patients are offered an opportunity to participate in this study, they will receive a single hyperbaric oxygen session. During the first session, hyperbaric oxygen will be administered at 3.0 atmospheres absolute (atm abs) for 25 minutes breathing oxygen, 5 minutes air breathing, 25 minutes oxygen breathing, 5 minutes air breathing, pressure reduced to 2.0 atm abs for 30 minutes breathing oxygen, 5 minutes air breathing, and 30 minutes oxygen breathing.
  For the second and third hyperbaric oxygen sessions, the subject will breathe 100% oxygen delivered at 2 atm abs for 90 minutes with two 5-minute air breathing periods.
  Other Names: Hyperbaric Oxygen; HBO2; HBO; HBOT
  Arms: Hyperbaric Oxygen (HBO2) - 3 sessions
Combination Product: Hyperbaric Oxygen (HBO2) - 1 session — During the first session, hyperbaric oxygen will be administered at 3.0 atmospheres absolute (atm abs) for 25 minutes breathing oxygen, 5 minutes air breathing, 25 minutes oxygen breathing, 5 minutes air breathing, pressure reduced to 2.0 atm abs for 30 minutes breathing oxygen, 5 minutes air breathing, and 30 minutes oxygen breathing.
  The second and third chamber sessions are sham sessions: room air delivered at 1.0 atmospheres absolute for 90 minutes with two sham 5-minute air breathing periods.
  Other Names: HBO2
  Arms: Hyperbaric Oxygen (HBO2) - 1 session

SUMMARY:
This randomized trial will investigate important clinical outcomes of patients with acute carbon monoxide poisoning randomized to receive either one or three hyperbaric oxygen treatments.

DETAILED DESCRIPTION:
All patients presenting with acute carbon monoxide poisoning will receive one hyperbaric oxygen treatment (barring contraindications for hyperbaric oxygen therapy). After this treatment, eligible patients who provide consent will be randomly allocated to receive two sham sessions, or two additional hyperbaric oxygen sessions administered in a double-blind fashion.

Outcome measures will be administered at 6 weeks and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic CO poisoning (headache, nausea, vomiting, dizziness, fatigue, muscle aches, slowed mentation, confusion, or loss of consciousness).
* Carboxyhemoglobin (COHb) levels > 10% or confirmation of poisoning with ambient levels > 50 ppm in a patient with symptoms compatible with CO poisoning and no other reasonable explanation for their signs and symptoms.
* Less than 24 hours from removal from the source of CO exposure and study enrollment.
* Accidental poisoning

Exclusion Criteria:

* Pregnancy
* Age < 18 years or > 79 years
* Complication during first hyperbaric oxygen session precluding subsequent hyperbaric oxygen.
* Intentional CO poisoning
* Unable to obtain informed consent
* Moribund patient
* Concomitant smoke inhalation with cyanide poisoning
* Bleomycin use within two weeks of study enrollment
* Intracardiac defibrillator that cannot be deactivated
* Non-English speaking
* Unlikely to return at 6 weeks
* History of central nervous system (CNS) disease (i.e., Alzheimer's, Parkinson's, dementia, demyelinating disease (MS), etc.)
* History of prior brain injury (i.e., stroke, traumatic brain injury)
* Presence of chronic debilitating disease likely to result in death within 12 months (i.e., kidney failure on dialysis, heart failure)
* Subject has a significant medical condition or conditions that would interfere with the treatment, safety, or compliance with the protocol.
* Intubated subjects
* Subjects requiring greater than 50% oxygen by non-rebreather facemask or exhibiting evidence of respiratory compromise or heart failure
* Subjects who, in the opinion of the investigator, are unable to comply with the requirements of the study or are unsuitable for any reason. The investigator and the Sponsor, prior to enrolling the subject on a case-by-case basis, must approve and document any waiver of these inclusion and exclusion criteria.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-06-03 (Actual); Primary Completion 2016-09-10 (Actual); Study Completion 2017-01-28 (Actual)

PRIMARY OUTCOMES:
6-week cognitive sequelae | 6 weeks after poisoning
  Presence of cognitive sequelae at 6-week follow-up

SECONDARY OUTCOMES:
Neurological examination | 6 weeks and 6 months after poisoning
  Presence of neurological abnormalities
Depression, anxiety or post-traumatic stress syndrome | 6 weeks and 6 months after poisoning
  Presence of depression, anxiety, or PTSD symptoms
Vocational assessment | 6 weeks and 6 months after poisoning
  Results of vocational testing
Patient self-reports of CO-related problems | 6 weeks and 6 months
  Participant-reported outcome

CONTACTS AND LOCATIONS:
Overall Officials: Lindell K Weaver, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (2):
- United States (2):
  - Intermountain LDS Hospital, Salt Lake City, Utah
  - Intermountain Medical Center, Salt Lake City, Utah

REFERENCES:
- [Background] Weaver LK, Hopkins RO, Chan KJ, Churchill S, Elliott CG, Clemmer TP, Orme JF Jr, Thomas FO, Morris AH. Hyperbaric oxygen for acute carbon monoxide poisoning. N Engl J Med. 2002 Oct 3;347(14):1057-67. doi: 10.1056/NEJMoa013121. PMID 12362006